CLINICAL TRIAL: NCT00871871
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Part Study to Evaluate the Multiple Dose Effects of Hydrochlorothiazide and Isosorbide Mononitrate on Glucose Homeostasis in Obese Patients With Hypertension
Brief Title: Multiple Dose Effects of Hydrochlorothiazide and Isosorbide Mononitrate on Glucose Homeostasis (MK-0000-117)(Completed)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-117; 2009_567
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2011-09-22 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part I, Placebo-HCTZ (Experimental): Placebo in Period 1 followed by HCTZ in Period 2
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Comparator: Placebo to HCTZ
- Part I, HCTZ-Placebo (Experimental): HCTZ in Period 1, followed by placebo in Period 2
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Comparator: Placebo to HCTZ
- Part II, Placebo-ISMN (Experimental): Placebo in Period 1, followed by ISMN in Period 2
  Interventions: Drug: Isosorbide mononitrate (ISMN); Drug: Comparator: Placebo to ISMN
- Part II, ISMN-Placebo (Experimental): ISMN in Period 1, followed by placebo in Period 2
  Interventions: Drug: Isosorbide mononitrate (ISMN); Drug: Comparator: Placebo to ISMN

INTERVENTIONS:
Drug: Hydrochlorothiazide (HCTZ) — HCTZ 50 mg (two 25 mg capsules) once daily for 4 weeks per treatment period.
  Other Names: HCTZ
  Arms: Part I, HCTZ-Placebo; Part I, Placebo-HCTZ
Drug: Comparator: Placebo to HCTZ — Placebo to HCTZ two 0 mg capsules once daily for 4 weeks per treatment period
  Arms: Part I, HCTZ-Placebo; Part I, Placebo-HCTZ
Drug: Isosorbide mononitrate (ISMN) — ISMN 60 mg extended release capsule once daily for 4 weeks per treatment period
  Arms: Part II, ISMN-Placebo; Part II, Placebo-ISMN
Drug: Comparator: Placebo to ISMN — Placebo to ISMN 0 mg capsule once daily for 4 weeks per treatment period
  Arms: Part II, ISMN-Placebo; Part II, Placebo-ISMN

SUMMARY:
This study will measure and compare changes in insulin production and sensitivity using the hyperglycemic clamp technique in obese patients with impaired glucose tolerance and hypertension treated with placebo, isosorbide mononitrate (ISMN) or hydrochlorothiazide (HCTZ).

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be post-menopausal
* Body Mass Index (BMI) of at least 29 kg/m^2
* Weight has been stable over the past 3 months
* Has never been treated for hypertension or is diagnosed with hypertension taking up to 2 anti-hypertensive medications
* Willing to stop hypertension treatment for 14 days prior to randomization and throughout the study
* Does not have a history of diabetes
* In good health with the exception of hypertension
* No history of abnormal heart rhythms
* Part I only: willing to comply with high potassium/low sodium diet for the duration of the study
* Willing to avoid strenuous physical activity during the study
* Nonsmoker and/or has not used nicotine for at least 3 months and agrees to refrain from use of tobacco-containing products throughout the study
* Agrees to refrain from consuming alcohol and caffeine during in-patient periods and to limit consumption at all other times during the study
* Agrees not to consume grapefruit, grapefruit products, and citrus, apple, and pineapple juices 2 weeks prior to administration of the first dose of study drug

Exclusion Criteria:

* History of any illness that may make their participation in the study unsafe or confuse the study results
* Taking spironolactone or eplerenone
* Cannot refrain from using any prescription or non-prescription drugs during the study
* On a weight loss program and is not in the maintenance phase
* Started a weight loss drug within 8 weeks of the first study visit
* Consumes excessive amounts of alcohol or caffeine
* Has had major surgery, donated or lost 1 unit of blood within 4 weeks of the first study visit
* History of multiple and/or severe allergies to drugs or food
* Is dehydrated

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants were place into two periods. 36 Part I participants received Hydrochlorothiazide (HCTZ) first, then placebo or placebo first, then HCTZ. A new group of 28 Part II participants received Isosorbide Mononitrate (ISMN) first, then placebo or placebo first, then ISMN.
Groups:
- HCTZ First, Then HCTZ Placebo; HCTZ Placebo First, Then HCTZ: Part I Overall: Placebo in Period 1 followed by hydrochlorothiazide (HCTZ) in Period 2 or HCTZ in Period 1, followed by placebo in Period 2
- ISMN First, Then ISMN Placebo; ISMN Placebo First, Then ISMN: Part II Overall: Placebo in Period 1, followed by isosorbide mononitrate (ISMN) in Period 2 or ISMN in Period 1, followed by placebo in Period 2
Period: Part I
Arm/Group | HCTZ First, Then HCTZ Placebo | HCTZ Placebo First, Then HCTZ | ISMN First, Then ISMN Placebo | ISMN Placebo First, Then ISMN
Started | 18 | 18 | 0 | 0
Completed | 15 | 15 | 0 | 0
Not Completed | 3 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — Laboratory abnormality | 0 | 1 | 0 | 0
Period: Part II
Arm/Group | HCTZ First, Then HCTZ Placebo | HCTZ Placebo First, Then HCTZ | ISMN First, Then ISMN Placebo | ISMN Placebo First, Then ISMN
Started | 0 | 0 | 13 | 15
Completed | 0 | 0 | 9 | 11
Not Completed | 0 | 0 | 4 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Part I Participants: Part I Overall: Hydrochlorothiazide (HCTZ) in Period 1 followed by Placebo in Period 2 or Placebo in Period 1, followed by HCTZ in Period 2
- All Part II Participants: Part II Overall: Isosorbide mononitrate (ISMN)in Period 1, followed by placebo in Period 2 or placebo in Period 1, followed by ISMN in Period 2
- Total: Total of all reporting groups
Arm/Group | All Part I Participants | All Part II Participants | Total
Number analyzed (Participants) | 36 | 28 | 64
Age, Continuous [Mean (Full Range); unit: years] | 57 [35 to 72] | 54 [37 to 73] | 55 [35 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Part I: Change in Insulin Secretion at Steady-state Compared to Placebo in Participants With Impaired Glucose Tolerance (IGT)
Description: Steady state was defined as 90-120 minutes post-dose. IGT was defined as a 2 hour plasma glucose >= 140 and <= 199 mg/dL during a 75g oral glucose tolerance test at screening.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants with IGT.
Measure: Least Squares Mean (Standard Deviation); unit: ng/minute
Groups:
- Hydrochlorothiazide (HCTZ): Part I: Participants on HCTZ in either Period 1 or Period 2
- Hydrochlorothiazide (HCTZ) Placebo: Part I: Participants on HCTZ Placebo in either Period 1 or Period 2
Arm/Group | Hydrochlorothiazide (HCTZ) | Hydrochlorothiazide (HCTZ) Placebo
Number analyzed (Participants) | 5 | 5
ng/minute | 3.44 (1.03) | 3.55 (1.03)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCTZ) vs Hydrochlorothiazide (HCTZ) Placebo; Test type: Superiority or Other; p = 0.067, ANCOVA — one-sided, alpha = 0.05; Least squares mean difference = -0.10, 90% CI 2-sided [-0.22 to 0.01]

2. Primary Outcome: Part I: Change in Insulin Secretion at Steady-state Compared to Placebo in Participants With Impaired Fasting Glucose (IFG)
Description: Steady state was defined as 90-120 minutes post-dose. IFG was defined as fasting plasma glucose (FPG) between 100 and 125 mg/dL at screening.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants with IFG.
Measure: Least Squares Mean (Standard Deviation); unit: ng/minute
Arm/Group | Hydrochlorothiazide (HCTZ) | Hydrochlorothiazide (HCTZ) Placebo
Number analyzed (Participants) | 7 | 8
ng/minute | 5.60 (1.45) | 4.50 (0.95)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCTZ) vs Hydrochlorothiazide (HCTZ) Placebo; Test type: Superiority or Other; p > 0.500, ANCOVA; Least squares mean difference = 1.10, 90% CI 2-sided [0.86 to 1.34]

3. Secondary Outcome: Part I: Change in the Ratio of Whole Body Glucose Disposal to Plasma Insulin at Steady State in Participants With Impaired Glucose Tolerant (IGT)
Description: Steady state was defined as 90-120 minutes post-dose. The ratio was the quantity of glucose disposed by the body per kg body weight per minute at steady state divided by the approximate steady state plasma insulin concentration. The approximate steady state plasma insulin concentration was estimated by the time-weighted average of the insulin concentration measured at 10 minute intervals in which time = 90, 100, 110, and 120 minutes. IGT was defined as a 2 hour plasma glucose >= 140 and <= 199 mg/dL during a 75g oral glucose tolerance test at screening.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants with IGT.
Measure: Least Squares Mean (Standard Deviation); unit: (mg/kg/minute)/(µIU/mL)
Arm/Group | Hydrochlorothiazide (HCTZ) | Hydrochlorothiazide (HCTZ) Placebo
Number analyzed (Participants) | 5 | 5
(mg/kg/minute)/(µIU/mL) | 0.061 (0.044) | 0.045 (0.041)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCTZ) vs Hydrochlorothiazide (HCTZ) Placebo; Test type: Superiority or Other; p = 0.130, ANOVA — one-sided, alpha = 0.05; Least squares mean difference = 0.016, 90% CI 2-sided [-0.012 to 0.044]

4. Primary Outcome: Part I: Change in Insulin Secretion at Steady-state Compared to Placebo in Participants Who Had Normal Glucose Tolerance (NGT)
Description: Steady state was defined as 90-120 minutes post-dose. NGT participants (FPG <100 mg/dL & 2 hour plasma glucose (PG) <140 mg/dL during a 75g oral glucose tolerance test (OGTT) at screening) were neither Impaired Glucose Tolerant (IGT) nor Impaired Fasting Glucose (IFG). IGT was defined as a 2 hour plasma glucose >= 140 and <= 199 mg/dL during a 75g oral glucose tolerance test at screening. IFG was defined as FPG between 100 and 125 mg/dL at screening.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants with NGT.
Measure: Least Squares Mean (Standard Deviation); unit: ng/minute
Arm/Group | Hydrochlorothiazide (HCTZ) | Hydrochlorothiazide (HCTZ) Placebo
Number analyzed (Participants) | 22 | 23
ng/minute | 5.54 (2.15) | 5.01 (1.63)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCTZ) vs Hydrochlorothiazide (HCTZ) Placebo; Test type: Superiority or Other; p > 0.500, ANCOVA; Least squares mean difference = 0.54, 90% CI 2-sided [0.40 to 0.67]

5. Primary Outcome: Part II: Ratio of Whole Body Glucose Disposal to Plasma Insulin at Steady-state
Description: Steady state was defined as 90-120 minutes post-dose. The ratio was the quantity of glucose disposed by the body per kg body weight per minute at steady state divided by the approximate steady state plasma insulin concentration. The approximate steady state plasma insulin concentration was estimated by the time-weighted average of the insulin concentration measured at 10 minute intervals in which time = 90, 100, 110, and 120 minutes.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants who took ISMN/placebo.
Measure: Least Squares Mean (Standard Deviation); unit: (mg/kg/minute)/(µIU/mL)
Groups:
- Isosorbide Mononitrate (ISMN): Part II: Participants on ISMN in either Period 1 or Period 2
- Isosorbide Mononitrate (ISMN) Placebo: Part II: Participants on ISMN Placebo in either Period 1 or Period 2
Arm/Group | Isosorbide Mononitrate (ISMN) | Isosorbide Mononitrate (ISMN) Placebo
Number analyzed (Participants) | 20 | 23
(mg/kg/minute)/(µIU/mL) | 0.040 (0.027) | 0.044 (0.041)
Statistical Analysis 1: Comparison: Isosorbide Mononitrate (ISMN) vs Isosorbide Mononitrate (ISMN) Placebo; Test type: Superiority or Other; p = 0.342, ANOVA — one-sided, alpha = 0.05; Least squares mean difference = 0.004, 90% CI 2-sided [-0.023 to 0.014]

6. Secondary Outcome: Part I: Change in the Ratio of Whole Body Glucose Disposal to Plasma Insulin at Steady State in Participants With Impaired Fasting Glucose (IFG)
Description: Steady state was defined as 90-120 minutes post-dose. The ratio was the quantity of glucose disposed by the body per kg body weight per minute at steady state divided by the approximate steady state plasma insulin concentration. The approximate steady state plasma insulin concentration was estimated by the time-weighted average of the insulin concentration measured at 10 minute intervals in which time = 90, 100, 110, and 120 minutes. IFG was defined as fasting plasma glucose (FPG) between 100 and 125 mg/dL at screening.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants with IFG.
Measure: Least Squares Mean (Standard Deviation); unit: (mg/kg/minute)/(µIU/mL)
Arm/Group | Hydrochlorothiazide (HCTZ) | Hydrochlorothiazide (HCTZ) Placebo
Number analyzed (Participants) | 7 | 8
(mg/kg/minute)/(µIU/mL) | 0.038 (0.019) | 0.037 (0.109)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCTZ) vs Hydrochlorothiazide (HCTZ) Placebo; Test type: Superiority or Other; p > 0.500, ANOVA; Least squares mean difference = 0.0016, 90% CI 2-sided [-0.008 to 0.011]

7. Secondary Outcome: Part I: Change in the Ratio of Whole Body Glucose Disposal to Plasma Insulin at Steady State in Participants With Normal Glucose Tolerant (NGT)
Description: Steady state was defined as 90-120 minutes post-dose. The ratio was the measure of the quantity of glucose disposed per unit of plasma insulin concentration (PIC). Approximate PIC was estimated by the time-weighted average of the insulin concentration measured at 10 minute intervals, time = 90, 100, 110, and 120 minutes. NGT participants (FPG <100 mg/dL & 2 hour PG <140 mg/dL during a 75g OGTT at screening) were neither IGT nor IFG at screening. IGT - defined as a 2 hour PG >= 140 and <= 199 mg/dL during a 75g OGTT at screening. IFG - defined as FPG between 100 and 125 mg/dL at screening.
Time Frame: 90 -120 minutes post-dose
Population: Number of participants with NGT.
Measure: Least Squares Mean (Standard Deviation); unit: (mg/kg/minute)/(µIU/mL)
Arm/Group | Hydrochlorothiazide (HCTZ) | Hydrochlorothiazide (HCTZ) Placebo
Number analyzed (Participants) | 22 | 23
(mg/kg/minute)/(µIU/mL) | 0.045 (0.028) | 0.042 (0.024)
Statistical Analysis 1: Comparison: Hydrochlorothiazide (HCTZ) vs Hydrochlorothiazide (HCTZ) Placebo; Test type: Superiority or Other; p > 0.500, ANOVA; Least squares mean difference = 0.003, 90% CI 2-sided [-0.003 to 0.010]

ADVERSE EVENTS:
Groups:
- HCTZ: Part I: Participants on HCTZ in either Period 1 or Period 2
- HCTZ Placebo: Part I: Participants on HCTZ Placebo in either Period 1 or Period 2
- ISMN: Part II: Participants on ISMN in either Period 1 or Period 2
- ISMN Placebo: Part II: Participants on ISMN Placebo in either Period 1 or Period 2
Arm/Group | HCTZ | HCTZ Placebo | ISMN | ISMN Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 29/36 | 25/36 | 26/28 | 17/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCTZ (N=36) | HCTZ Placebo (N=36) | ISMN (N=28) | ISMN Placebo (N=28)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 2 | 0 | 2
Blood potassium decreased (Investigations) | 4 | 0 | 0 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 3 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 4 | 2 | 3 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 11 | 12 | 26 | 14
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 5 | 0
Nocturia (Renal and urinary disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 4 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.